CLINICAL TRIAL: NCT01935440
Title: A Comprehensive Approach to Secondary HIV Prevention and Care Among Positives
Acronym: P&T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Carl Latkin, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01DA032217 (NIH); R01DA032217 (NIH)
Record Dates: First submitted 2013-08-20; First posted 2013-09-05 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: HIV
Keywords: HIV, drug use

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prevention & Testing Control (Active Comparator): The comparison condition is focused on basic HIV risk reduction , safety and preventing drug overdose.
  Interventions: Behavioral: Prevention & Testing Control
- Prevention & Testing Intervention (Experimental): The intervention condition is training on peer outreach skills which includes talking to HIV positive social network members about HIV care, medication adherence and HIV risk reduction.
  Interventions: Behavioral: Prevention & Testing

INTERVENTIONS:
Behavioral: Prevention & Testing — 6 group sessions, 1 individual session, and 1 dyad session
  Arms: Prevention & Testing Intervention
Behavioral: Prevention & Testing Control — 7 group sessions
  Arms: Prevention & Testing Control

SUMMARY:
The goal of this study is to conduct an HIV prevention intervention to train HIV seropositive drug users to be peer health educators.

DETAILED DESCRIPTION:
The primary objective of this funded research is to conduct an HIV prevention intervention to train HIV seropositive drug users to be peer health educators to: (1) recruit their high risk social network members for voluntary HIV counseling and testing (VCT) at the research clinic, (2) promote risk reduction among social network members, and (3) promote engagement in HIV care by encouraging HIV seropositive network members to schedule and keep HIV primary care appointments. There will be four types of participants in the Full Trial: 1) Index, 2) Testing Network 3) Longitudinal Network and 4) HIV positive network participants. This longitudinal study includes baseline, 6-months, and 12-month assessments

ELIGIBILITY:
Inclusion Criteria:

Index

1. 18 years old or older
2. documentation of HIV positive status
3. report one of following risk behaviors in past 90 days: sharing injection equipment, use of crack cocaine, or unprotected vaginal or anal sex

Testing network

1. 18 or older
2. provided testing coupon provided by an index participant

Longitudinal network participant-

1. tested HIV negative at the Lighthouse via redeeming a testing coupon
2. reported interacting with index who gave the coupon at least weekly
3. report one of following risk behaviors in the prior 90 days: sharing injection equipment, use of crack cocaine, or unprotected vaginal or anal sex

Positive Networks

1. HIV positive
2. report one of following risk behaviors in the prior 90 days: sharing injection equipment, use of crack cocaine, or unprotected vaginal or anal sex

Exclusion Criteria:

Index- already enrolled in the study as a Network participant

Testing network- already enrolled in the study as a Network participant

Longitudinal network- a) already enrolled in the study as a Network participant b) already enrolled in the study as a Index participant

Positive network- a) already enrolled in the study as a Network participant b) already enrolled in the study as a Index participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
change in HIV medication adherence | 6 month
change in frequency in attending HIV medical appointments | 6 month

SECONDARY OUTCOMES:
change in sharing injection equipment | 6 month
change in condom use | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Carl A Latkin, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Lighhouse Studies @ Peer Point, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided